CLINICAL TRIAL: NCT01969708
Title: Study of COmparative Treatments for REtinal Vein Occlusion 2 [SCORE2]: a Multicenter, Prospective, Randomized Non-inferiority Trial of Eyes With Macular Edema Secondary to Central Retinal Vein Occlusion, Comparing Intravitreal Bevacizumab Every 4 Weeks With Intravitreal Aflibercept Every 4 Weeks.
Brief Title: Study of Comparative Treatments for Retinal Vein Occlusion 2 (SCORE2)
Acronym: SCORE2
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: The Emmes Company, LLC (Industry)
Collaborators: National Eye Institute (NEI) (NIH); Milton S. Hershey Medical Center (Other); University of Wisconsin, Madison (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: SCORE2; U10EY023529 (NIH); U10EY023533 (NIH); U10EY023521 (NIH)
Record Dates: First submitted 2013-10-22; First posted 2013-10-25 (Estimated); Results first posted 2018-08-21 (Actual); Last update posted 2021-06-22 (Actual); Status verified 2021-06

CONDITIONS: Central Retinal Vein Occlusion
MeSH Terms: conditions — Retinal Vein Occlusion | interventions — aflibercept; Bevacizumab

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- aflibercept (Active Comparator): 2.0 mg aflibercept every 4 weeks
  Interventions: Drug: aflibercept
- bevacizumab (Active Comparator): 1.25 mg bevacizumab every 4 weeks
  Interventions: Drug: bevacizumab

INTERVENTIONS:
Drug: aflibercept
  Other Names: EYLEA
  Arms: aflibercept
Drug: bevacizumab
  Other Names: Avastin
  Arms: bevacizumab

SUMMARY:
SCORE2 is a multicenter, prospective, randomized, phase III clinical trial in which all participants enrolled will be followed for up to 2.5 years. SCORE2 is designed as a non-inferiority trial, with study eyes randomized to intravitreal bevacizumab (1.25 mg) every 4 weeks vs. intravitreal aflibercept (2.0 mg) every 4 weeks. SCORE2 aims to determine if bevacizumab is non-inferior to aflibercept for the treatment of macular edema associated with central retinal vein occlusion (CRVO), with the primary outcome of visual acuity measured at Month 6.

DETAILED DESCRIPTION:
The primary objective of SCORE2 is to test for non-inferiority based on mean change from baseline in visual acuity letter score at Month 6 for eyes randomized to intravitreal bevacizumab every 4 weeks compared with eyes randomized to intravitreal aflibercept every 4 weeks using a non-inferiority margin of 5 letters.

Secondary objectives of SCORE2 are to:

* compare the bevacizumab and the aflibercept groups with regards to central retinal thickness, as measured with spectral domain optical coherence tomography (SD-OCT), at Month 6 and change between baseline and Month 6;
* assess Month 12 visual acuity and SD-OCT outcomes associated with different dosing strategies after Month 6 in participants who respond well to treatment;
* assess Month 12 visual acuity and SD-OCT outcomes associated with alternative treatment strategies after Month 6 in participants who respond poorly to treatment;
* compare area of retinal ischemia and rates of neovascular complications of CRVO in the bevacizumab vs. aflibercept groups;
* add to our knowledge of the safety profile of these anti-vascular endothelial growth factor (VEGF) medications in the setting of eyes with macular edema secondary to CRVO;
* conduct a cost effectiveness analysis comparing intravitreal bevacizumab to intravitreal aflibercept to assess the economic implications from a payor perspective using decision analytic methods.

Other exploratory aims of SCORE2 are to:

* investigate the correlation of features identified through SD-OCT segmentation analysis, such as the inner segment-outer segment (IS-OS) junction (also known as the ellipsoid zone), with such characteristics as visual acuity and central retinal thickness;
* investigate the correlation of area of peripheral retinal nonperfusion from widefield fluorescein angiography with visual acuity and central retinal thickness, and the prognostic value of baseline peripheral and central retina perfusion status in predicting disease course and treatment responsiveness;
* investigate the correlation of features on adaptive optics imaging with such characteristics as visual acuity and central retinal thickness.

ELIGIBILITY:
Inclusion Criteria:

* Participants must have center-involved macular edema secondary to CRVO. Eyes may be enrolled as early as the time of diagnosis of the macular edema. The definition of CRVO used in SCORE will also be used for the purposes of SCORE2: a CRVO is defined as an eye that has retinal hemorrhage or other biomicroscopic evidence of retinal vein occlusion (e.g., telangiectatic capillary bed) and a dilated venous system (or previously dilated venous system) in all 4 quadrants.
* Due to the similarities of a hemiretinal vein occlusion (HRVO) to CRVO,HRVO will be classified as CRVO for the purposes of this clinical trial. Eyes classified as having a HRVO will be limited to no more than 25% of the planned sample size. A HRVO is defined as an eye that has retinal hemorrhage or other biomicroscopic evidence of retinal vein occlusion (e.g. telangiectatic capillary bed) and a dilated venous system (or previously dilated venous system) in 5 or more clock hours but less than all 4 quadrants. Typically, a HRVO is a retinal vein occlusion that involves 2 altitudinal quadrants.
* E-Early Treatment Diabetic Retinopathy Study (ETDRS)visual acuity score of greater than or equal to 19 letters (approximately 20/400) and less than or equal to 73 letters (approximately 20/40) by the ETDRS visual acuity protocol. The investigator must believe that a study eye with visual acuity between 19 and 33 letters is perfused.
* Retinal thickness on SD-OCT measurement, defined as central subfield thickness of 300 µm or greater. If the SD-OCT measurement is taken from a Heidelberg Spectralis Machine, the central subfield thickness should be 320 µm or greater.
* Media clarity, pupillary dilation and participant cooperation sufficient for adequate fundus photographs.

Exclusion Criteria:

* A condition that, in the opinion of the investigator, would preclude participation in the study (e.g., chronic alcoholism or drug abuse, personality disorder or use of major tranquilizers indicating difficulty in long term follow-up, likelihood of survival of less than 12 months).
* Participation in an investigational trial within 30 days of study entry that involved treatment with any drug that has not received regulatory approval at time of study entry.
* History of allergy to any anti-VEGF agent, corticosteroid, or component of the delivery vehicle.
* The participant will be moving out of the area of the clinical site to an area not covered by another clinical site during the 12 months of the study.
* Positive urine pregnancy test: all women of childbearing potential (those who are pre-menopausal and not surgically sterilized) may participate only if they have a negative urine pregnancy test, and if they do not intend to become pregnant during the timeframe of the study. Women who are sexually active with a male partner must agree to use at least one of the following birth control methods: hormonal therapy such as oral, implantable or injectable chemical contraceptives; mechanical therapy such as spermicide in conjunction with a barrier such as a condom or diaphragm; intrauterine device (IUD); or surgical sterilization of partner.
* Women who are breast-feeding.
* Examination evidence of vitreoretinal interface disease (e.g., vitreomacular traction, epiretinal membrane), either on clinical examination or OCT thought to be contributing to macular edema.
* An eye that, in the investigator's opinion, would not benefit from resolution of macular edema such as eyes with foveal atrophy, dense pigmentary changes or dense subfoveal hard exudates.
* Presence of an ocular condition that, in the opinion of the investigator, might affect macular edema or alter visual acuity during the course of the study (e.g., age-related macular degeneration, uveitis or other ocular inflammatory disease, neovascular glaucoma, iris neovascularization, Irvine-Gass Syndrome, prior macula-off rhegmatogenous retinal detachment).
* Presence of a substantial cataract that, in the opinion of the investigator, is likely to be decreasing visual acuity by 3 lines or more (i.e., a 20/40 cataract).
* History of laser photocoagulation for macular edema within 3 months prior to randomization.
* History of intravitreal corticosteroid within 4 months of randomization.
* Intravitreal anti-VEGF injection within 2 months of randomization. Note: Enrollment will be limited to no more than 25% of the planned sample size with any history of anti-VEGF treatment. Once this number of eyes has been enrolled, any history of anti-VEGF treatment will be an exclusion criterion. For enrollment of study eyes with prior intravitreal anti-VEGF agents, in the opinion of the investigator, the treatment response to prior anti-VEGF treatment must be either incomplete or the study eye had developed recurrent CRVO-associated macular edema, such that the study eye would benefit from additional anti-VEGF treatment.
* History of peribulbar or retrobulbar corticosteroid use for any reason within 2 months prior to randomization.
* History of panretinal scatter photocoagulation (PRP) or sector laser photocoagulation within 3 months prior to randomization or anticipated within the next 3 months following randomization.
* History of major ocular surgery (including cataract extraction, scleral buckle, any intraocular surgery, etc.) within 4 months prior to randomization or anticipated within the next 6 months following randomization.
* History of yttrium aluminum garnet (YAG) capsulotomy performed within 2 months prior to randomization.
* Aphakia.
* Presence of an anterior chamber intraocular lens
* Examination evidence of external ocular infection, including conjunctivitis, chalazion or significant blepharitis.
* History of macular detachment.
* Examination evidence of any diabetic retinopathy.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 362 (Actual)
Dates: Start 2014-09 (Actual); Primary Completion 2016-11 (Actual); Study Completion 2021-03 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Ingrid U Scott, M.D., M.P.H., Study Chair — Penn State College of Medicine
Locations (72):
- United States (72):
  - Retinal Consultants of AZ, Phoenix, Arizona
  - Retina Centers, P.C., Tucson, Arizona
  - Northern California Retina Vitreous Associates, Mountain View, California
  - East Bay Retina Consultants, Inc., Oakland, California
  - Southern California Desert Retina Consultants, Palm Desert, California
  - University of California Davis, Medical Center, Sacramento, California
  - Retinal Consultants Medical Group, Inc., Sacramento, California
  - University of California, San Francisco, San Francisco, California
  - New England Retina Associates, New London, Connecticut
  - Retina Group of Florida, Fort Lauderdale, Florida
  - National Ophthalmic Research Institute, Fort Myers, Florida
  - University of Florida, Dept of Ophthalmology, Jacksonville, Florida
  - Florida Retina Consultants, Lakeland, Florida
  - Sarasota Retina Institute, Sarasota, Florida
  - Center for Retina and Macular Disease, Winter Haven, Florida
  - Florida Retina Consultants, Winter Haven, Florida
  - Emory University Eye Center, Atlanta, Georgia
  - Southeast Retina Center, Augusta, Georgia
  - Georgia Retina, P.C., Marietta, Georgia
  - Illinois Eye and Ear Infirmary UIC Dept. of Ophthalmology, Chicago, Illinois
  - Thomas A. Ciulla, MD, PC, Indianapolis, Indiana
  - Sabates Eye Centers, Leawood, Kansas
  - Retina Associates, PA, Shawnee Mission, Kansas
  - Retina Associates of Kentucky, Lexington, Kentucky
  - University of Kentucky, Lexington, Kentucky
  - Paducah Retinal Center, Paducah, Kentucky
  - Elman Retina Group, PA, Baltimore, Maryland
  - The Retina Group of Washington, Chevy Chase, Maryland
  - Elman Retina Group, P.A., Glen Burnie, Maryland
  - Cumberland Valley Retina Consultants, Hagerstown, Maryland
  - Elman Retina Group, P.A., Pikesville, Maryland
  - Henry Ford Health System, Detroit, Michigan
  - TLC Eyecare & Laser Centers, Jackson, Michigan
  - VitreoRetinal Surgery, Minneapolis, Minnesota
  - Mayo Clinic, Rochester, Minnesota
  - The Retina Institute, St Louis, Missouri
  - UNMC Truhlsen Eye Institute, Omaha, Nebraska
  - Retina Consultants of Nevada, Las Vegas, Nevada
  - Delaware Valley Retina Associates, Lawrenceville, New Jersey
  - NJ Retina, New Brunswick, New Jersey
  - New York Eye and Ear Infirmary, New York, New York
  - Retina Associates of Western New York, Rochester, New York
  - University of Rochester Flaum Eye Institute, Rochester, New York
  - Retina Vitreous Surgeon of CNY, PC, Syracuse, New York
  - Charlotte Eye Ear Nose & Throat Associates, P.A., Charlotte, North Carolina
  - Charlotte Eye Ear Nose & Throat Associates, P.A., Statesville, North Carolina
  - Retina Associates of Cleveland, Inc., Cleveland, Ohio
  - The Ohio State University, Columbus, Ohio
  - Dean McGee Eye Institute, Oklahoma City, Oklahoma
  - Retina Northwest, PC, Portland, Oregon
  - Casey Eye Institute / OHSU, Portland, Oregon
  - Retina Vitreous Consultants, Monroeville, Pennsylvania
  - Scheie Eye Institute, Philadelphia, Pennsylvania
  - Carolinas Centers for Sight, PC, Florence, South Carolina
  - Palmetto Retina Center, West Columbia, South Carolina
  - Black Hills Regional Eye Institute, Rapid City, South Dakota
  - Southeastern Retina Associates, PC, Knoxville, Tennessee
  - Tennessee Retina, PC, Nashville, Tennessee
  - Vanderbilt Eye Institute, Nashville, Tennessee
  - Retina Research Institute of Texas, Abilene, Texas
  - Texas Retina Associates, Arlington, Texas
  - The Retina Research Center, Austin, Texas
  - Texas Retina Associates, Dallas, Texas
  - Charlotte Eye Ear Nose & Throat Associates, P.A., Houston, Texas
  - Retina & Vitreous of Texas, Houston, Texas
  - Retina Consultants of Houston, PA, Houston, Texas
  - Valley Retina Institute, PA, McAllen, Texas
  - Medical Center Ophthalmology Associates, San Antonio, Texas
  - Retinal Consultants of San Antonio, San Antonio, Texas
  - The Retina Group of Washington, Fairfax, Virginia
  - University of Wisconsin, Madison, Wisconsin
  - Medical College of Wisconsin, Milwaukee, Wisconsin

IPD SHARING:
Plan to Share IPD: Yes
SCORE2 will follow specific plans for sharing of research data. After analysis, the final data set can be provided after appropriate procedures are implemented to preserve the anonymity of the records, specifically where protected health information (PHI) is required. Upon request, anonymized data will be shared under confidentiality agreements with researchers interested in the project.
Time Frame: The time frame will be determined
Access Criteria: Confidentiality agreements will be required before anonymized data will be shared.

REFERENCES:
- [Background] Scott IU, VanVeldhuisen PC, Ip MS, Blodi BA, Oden NL, Figueroa M; SCORE2 Investigator Group. SCORE2 Report 1: Techniques to Optimize Recruitment in Phase III Clinical Trials of Patients With Central Retinal Vein Occlusion. Am J Ophthalmol. 2016 Oct;170:25-31. doi: 10.1016/j.ajo.2016.07.011. Epub 2016 Jul 19. PMID 27450625
- [Background] Scott IU, VanVeldhuisen PC, Ip MS, Blodi BA, Oden NL, Figueroa M, Dugel PU; SCORE2 Investigator Group. SCORE2 Report 2: Study Design and Baseline Characteristics. Ophthalmology. 2017 Feb;124(2):245-256. doi: 10.1016/j.ophtha.2016.09.038. Epub 2016 Nov 15. PMID 27863843
- [Background] Scott IU, VanVeldhuisen PC, Ip MS, Blodi BA, Oden NL, King J, Antoszyk AN, Peters MA, Tolentino M; SCORE2 Investigator Group. Baseline Factors Associated With 6-Month Visual Acuity and Retinal Thickness Outcomes in Patients With Macular Edema Secondary to Central Retinal Vein Occlusion or Hemiretinal Vein Occlusion: SCORE2 Study Report 4. JAMA Ophthalmol. 2017 Jun 1;135(6):639-649. doi: 10.1001/jamaophthalmol.2017.1141. PMID 28492860
- [Background] Scott IU, Figueroa MJ, Oden NL, Ip MS, Blodi BA, VanVeldhuisen PC; SCORE2 Investigator Group. SCORE2 Report 5: Vision-Related Function in Patients With Macular Edema Secondary to Central Retinal or Hemiretinal Vein Occlusion. Am J Ophthalmol. 2017 Dec;184:147-156. doi: 10.1016/j.ajo.2017.10.008. Epub 2017 Oct 23. PMID 29074161
- [Background] Scott IU, VanVeldhuisen PC, Ip MS, Blodi BA, Oden NL, Altaweel M, Berinstein DM; SCORE2 Investigator Group. Comparison of Monthly vs Treat-and-Extend Regimens for Individuals With Macular Edema Who Respond Well to Anti-Vascular Endothelial Growth Factor Medications: Secondary Outcomes From the SCORE2 Randomized Clinical Trial. JAMA Ophthalmol. 2018 Apr 1;136(4):337-345. doi: 10.1001/jamaophthalmol.2017.6843. PMID 29476687
- [Background] Peterson JS, Rockwell K Jr, Scott IU, Ip MS, VanVeldhuisen PC, Blodi BA; SCORE2 Investigator Group. LONG-TERM PHYSICAL STABILITY, STERILITY, AND ANTI-VEGF BIOACTIVITY OF REPACKAGED BEVACIZUMAB IN 2-ML GLASS VIALS. Retina. 2019 Sep;39(9):1802-1809. doi: 10.1097/IAE.0000000000002212. PMID 29746405
- [Background] Ip MS, Oden NL, Scott IU, VanVeldhuisen PC, Blodi BA, Ghuman T, Baker CW; SCORE2 Investigator Group. Month 12 Outcomes After Treatment Change at Month 6 Among Poor Responders to Aflibercept or Bevacizumab in Eyes With Macular Edema Secondary to Central or Hemiretinal Vein Occlusion: A Secondary Analysis of the SCORE2 Study. JAMA Ophthalmol. 2019 Mar 1;137(3):281-287. doi: 10.1001/jamaophthalmol.2018.6111. PMID 30589922
- [Background] Etheridge T, Dobson ETA, Wiedenmann M, Papudesu C, Scott IU, Ip MS, Eliceiri KW, Blodi BA, Domalpally A. A semi-automated machine-learning based workflow for ellipsoid zone analysis in eyes with macular edema: SCORE2 pilot study. PLoS One. 2020 Apr 30;15(4):e0232494. doi: 10.1371/journal.pone.0232494. eCollection 2020. PMID 32353052
- [Background] Hendrick A, VanVeldhuisen PC, Scott IU, King J, Blodi BA, Ip MS, Khurana RN, Oden NL; SCORE2 Investigator Group. SCORE2 Report 13: Intraretinal Hemorrhage Changes in Eyes With Central or Hemiretinal Vein Occlusion Managed With Aflibercept, Bevacizumab or Observation. Secondary Analysis of the SCORE and SCORE2 Clinical Trials. Am J Ophthalmol. 2021 Feb;222:185-193. doi: 10.1016/j.ajo.2020.08.030. Epub 2020 Aug 20. PMID 32828880
- [Background] Etheridge T, Dobson ETA, Wiedenmann M, Oden N, VanVeldhuisen P, Scott IU, Ip MS, Eliceiri KW, Blodi BA, Domalpally A. Ellipsoid Zone Defects in Retinal Vein Occlusion Correlates With Visual Acuity Prognosis: SCORE2 Report 14. Transl Vis Sci Technol. 2021 Mar 1;10(3):31. doi: 10.1167/tvst.10.3.31. PMID 34003964
- [Background] Etheridge T, Blodi B, Oden N, Van Veldhuisen P, Scott IU, Ip MS, Mititelu M, Domalpally A. Spectral Domain OCT Predictors of Visual Acuity in the Study of COmparative Treatments for REtinal Vein Occlusion 2: SCORE 2 Report 15. Ophthalmol Retina. 2021 Oct;5(10):991-998. doi: 10.1016/j.oret.2020.12.016. Epub 2020 Dec 26. PMID 33373715
- [Result] Scott IU, VanVeldhuisen PC, Ip MS, Blodi BA, Oden NL, Awh CC, Kunimoto DY, Marcus DM, Wroblewski JJ, King J; SCORE2 Investigator Group. Effect of Bevacizumab vs Aflibercept on Visual Acuity Among Patients With Macular Edema Due to Central Retinal Vein Occlusion: The SCORE2 Randomized Clinical Trial. JAMA. 2017 May 23;317(20):2072-2087. doi: 10.1001/jama.2017.4568. PMID 28492910
- [Derived] Aref AA, Scott IU, Oden NL, Ip MS, VanVeldhuisen PC, Blodi BA; SCORE and SCORE2 Study Investigator Groups. Intraocular Pressure in Eyes With Retinal Vein Occlusion Compared With Fellow Eyes: Study of Comparative Treatments for Retinal Vein Occlusion 2 (SCORE2) Report 27. JAMA Ophthalmol. 2023 Dec 1;141(12):1172-1174. doi: 10.1001/jamaophthalmol.2023.5159. PMID 37943541
- [Derived] Scott IU, Oden NL, VanVeldhuisen PC, Ip MS, Blodi BA; SCORE2 Investigator Group. SCORE2 Report 24: Nonlinear Relationship of Retinal Thickness and Visual Acuity in Central Retinal and Hemiretinal Vein Occlusion. Ophthalmology. 2023 Oct;130(10):1066-1072. doi: 10.1016/j.ophtha.2023.05.023. Epub 2023 May 21. PMID 37220815
- [Derived] Scott IU, Oden NL, VanVeldhuisen PC, Ip MS, Blodi BA; SCORE2 Investigator Group. SCORE2 Report 20: Relationship of Treatment Discontinuation With Visual Acuity and Central Subfield Thickness Outcomes. Am J Ophthalmol. 2023 Apr;248:157-163. doi: 10.1016/j.ajo.2022.12.026. Epub 2022 Dec 28. PMID 36584835
- [Derived] Scott IU, VanVeldhuisen PC, Oden NL, Ip MS, Blodi BA; SCORE2 Investigator Group. Month 60 Outcomes After Treatment Initiation With Anti-Vascular Endothelial Growth Factor Therapy for Macular Edema Due to Central Retinal or Hemiretinal Vein Occlusion. Am J Ophthalmol. 2022 Aug;240:330-341. doi: 10.1016/j.ajo.2022.04.001. Epub 2022 Apr 21. PMID 35461831
- [Derived] Aref AA, Scott IU, VanVeldhuisen PC, King J, Ip MS, Blodi BA, Oden NL; Study of Comparative Treatments for Retinal Vein Occlusion 2 (SCORE2) Investigator Group. Intraocular Pressure-Related Events After Anti-Vascular Endothelial Growth Factor Therapy for Macular Edema Due to Central Retinal Vein Occlusion or Hemiretinal Vein Occlusion: SCORE2 Report 16 on a Secondary Analysis of a Randomized Clinical Trial. JAMA Ophthalmol. 2021 Dec 1;139(12):1285-1291. doi: 10.1001/jamaophthalmol.2021.4395. PMID 34709363
- [Derived] Khurana RN, Oden NL, VanVeldhuisen PC, Scott IU, Blodi BA, Ip MS; SCORE2 Investigator Group. Association between early and late response in eyes with central or hemiretinal vein occlusion treated with anti-VEGF agents : SCORE2 report 12: secondary analysis of the SCORE2 clinical trial. Graefes Arch Clin Exp Ophthalmol. 2021 Jul;259(7):1839-1851. doi: 10.1007/s00417-020-05018-7. Epub 2021 Jan 7. PMID 33415354
- [Derived] Scott IU, Oden NL, VanVeldhuisen PC, Ip MS, Blodi BA, Chan CK; SCORE2 Investigator Group. Month 24 Outcomes After Treatment Initiation With Anti-Vascular Endothelial Growth Factor Therapy for Macular Edema Due to Central Retinal or Hemiretinal Vein Occlusion: SCORE2 Report 10: A Secondary Analysis of the SCORE2 Randomized Clinical Trial. JAMA Ophthalmol. 2019 Dec 1;137(12):1389-1398. doi: 10.1001/jamaophthalmol.2019.3947. PMID 31600368
- [Derived] Scott IU, VanVeldhuisen PC, Barton F, Oden NL, Ip MS, Blodi BA, Worrall M, Fish GE; Study of Comparative Treatments for Retinal Vein Occlusion 2 Investigator Group. Patient-Reported Visual Function Outcomes After Anti-Vascular Endothelial Growth Factor Therapy for Macular Edema Due to Central Retinal or Hemiretinal Vein Occlusion: Preplanned Secondary Analysis of a Randomized Clinical Trial. JAMA Ophthalmol. 2019 Aug 1;137(8):932-938. doi: 10.1001/jamaophthalmol.2019.1519. PMID 31169862
- Available data/document: Study Protocol: PB2016-103333 — https://ntrl.ntis.gov/NTRL/ — SCORE2 Protocol Version 3.0 (the Identifier for the appendices is PB2016-103334)

RESULTS

PARTICIPANT FLOW:
Recruitment Details: The SCORE2 randomized noninferiority clinical trial was conducted at 66 private practice or academic centers in the United States, and included 362 patients with macular edema due to central retinal or hemiretinal vein occlusion who were randomized 1:1 to receive aflibercept or bevacizumab.
Pre-assignment Details: Participants were assigned to a treatment arm at enrollment.
Groups:
- Aflibercept: 2.0 mg aflibercept every 4 weeks
  aflibercept
- Bevacizumab: 1.25 mg bevacizumab every 4 weeks
  bevacizumab
Period: Overall Study
Arm/Group | Aflibercept | Bevacizumab
Started | 180 | 182
Completed | 175 | 173
Not Completed | 5 | 9

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Aflibercept | Bevacizumab | Total
Number analyzed (Participants) | 180 | 182 | 362
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 67 | 67 | 134
  >=65 years | 113 | 115 | 228
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 82 | 75 | 157
  Male | 98 | 107 | 205
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 16 | 22 | 38
  Not Hispanic or Latino | 164 | 160 | 324
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 8 | 2 | 10
  Asian | 4 | 2 | 6
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 28 | 26 | 54
  White | 132 | 146 | 278
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 8 | 6 | 14
Region of Enrollment [Number; unit: participants]
  United States | 180 | 182 | 362
Visual Acuity Letter Score (VALS) of Study Eye [Mean (Standard Deviation); unit: letters read] — The participant is refracted for best corrected vision, and then reads single letters on an electronic visual acuity tester at a 3 meter distance according to a specific algorithm. A letter score is provided that ranges from 0 (unable to ready any letters) to 100. A visual acuity letter score of 85 corresponds to a visual acuity of 20/20 as a Snellen equivalent.
  letters read | 50.3 (15.2) | 50.4 (15.3) | 50.3 (15.2)
Time between diagnosis of macular edema and randomization [Mean (Standard Deviation); unit: months] | 8 (17) | 5 (10) | 7 (14)
Spectral Domain-Optical Coherence Tomography (SD-OCT) central subfield thickness [Mean (Standard Deviation); unit: um] | 652.4 (214.6) | 678.2 (233.3) | 665.5 (224.4)
Prior anti-vascular endothelial growth factor (VEGF) treatment [Count of Participants; unit: Participants] | 65 | 56 | 121
Prior intravitreal steroid use [Count of Participants; unit: Participants] | 16 | 12 | 28
Hemiretinal vein occlusion [Count of Participants; unit: Participants] | 26 | 31 | 57
Cataract extraction [Count of Participants; unit: Participants] | 43 | 55 | 98
History of cataract [Count of Participants; unit: Participants] | 108 | 95 | 203
Diabetes mellitus type 1 [Count of Participants; unit: Participants] | 1 | 0 | 1
Diabetes mellitus type 2 [Count of Participants; unit: Participants] | 54 | 59 | 113
Hypertensive [Count of Participants; unit: Participants] | 140 | 138 | 278
Coronary artery disease [Count of Participants; unit: Participants] | 26 | 30 | 56
National Eye Institute (NEI) Visual Function Questionnaire (VFQ)-25 overall score [Mean (Standard Deviation); unit: total score] — For the National Eye Institute (NEI) Visual Function Questionnaire (VFQ)-25, respondents answer a series of multiple-choice questions about their vision and how it affects daily life. The overall scores range from 0 to 100, with higher scores representing better functioning.
  total score | 77 (15) | 77 (17) | 77 (16)

OUTCOME MEASURES:

1. Primary Outcome: Mean Change From Baseline in Best-corrected Early Treatment Diabetic Retinopathy Study (ETDRS) Visual Acuity Letter Score at Month 6
Description: The primary analysis is based on observed data at 6 months. The measure is calculated by subtracting the baseline visual acuity letter score from the month 6 visual acuity letter score. The participant is refracted for best corrected vision, and then reads single letters on an electronic visual acuity tester at a 3 meter distance according to a specific algorithm. A letter score is provided that ranges from 0 (unable to ready any letters) to 100. A visual acuity letter score of 85 corresponds to a visual acuity of 20/20 as a Snellen equivalent.
Time Frame: Month 0 to 6
Population: All participants with visual acuity letter score recorded at Month 6
Measure: Mean (95% Confidence Interval); unit: letters read
Arm/Group | Aflibercept | Bevacizumab
Number analyzed (Participants) | 175 | 173
letters read | 18.9 [16.62 to 21.15] | 18.6 [16.16 to 21.09]

2. Secondary Outcome: Number of Study Eyes With Gain of ≥15 Letters in Visual Acuity Letter Score at Month 6
Description: The measure is the number of study eyes that gained at least 15 letters in their visual acuity letter score at month 6
Time Frame: Month 0 to 6
Population: All participants with visual acuity letter score recorded at Month 6
Measure: Number; unit: study eyes
Arm/Group | Aflibercept | Bevacizumab
Number analyzed (Participants) | 175 | 173
study eyes | 114 | 106

3. Secondary Outcome: Number of Study Eyes With Visual Acuity Letter Score of 70 or Better at Month 6
Description: The measure is the number of study eyes with a visual acuity letter score of 70 (Snellen equivalent of 20/40) or better at month 6
Time Frame: Month 0 to 6
Population: All participants with visual acuity letter score recorded at Month 6
Measure: Number; unit: study eyes
Arm/Group | Aflibercept | Bevacizumab
Number analyzed (Participants) | 175 | 173
study eyes | 101 | 99

4. Secondary Outcome: Mean Spectral-domain Optical Coherence Tomography Central Subfield Thickness
Description: The measure is the mean central subfield thickness at month 6 measured by spectral-domain optical coherence tomography
Time Frame: Month 0 to 6
Population: All participants with central subfield thickness recorded at baseline and Month 6
Measure: Mean (95% Confidence Interval); unit: um
Arm/Group | Aflibercept | Bevacizumab
Number analyzed (Participants) | 164 | 171
um | 231.3 [220.8 to 241.8] | 287.9 [269.4 to 306.4]

5. Secondary Outcome: Mean Change From Baseline in Spectral Domain Optical Coherence Tomography Central Subfield Thickness at Month 6
Description: The measure is calculated by subtracting the baseline central subfield thickness from the month 6 central subfield thickness
Time Frame: Month 0 to 6
Population: All participants with central subfield thickness recorded at baseline and Month 6
Measure: Mean (95% Confidence Interval); unit: um
Arm/Group | Aflibercept | Bevacizumab
Number analyzed (Participants) | 164 | 171
um | -425 [-461 to -389] | -387 [-426 to -348]

6. Secondary Outcome: Number of Study Eyes With Central Subfield Thickness <300 μm, no Subretinal Fluid, no Intraretinal Fluid, and no Cystoid Spaces
Description: The measure is the number of study eyes with central subfield thickness <300 μm, no subretinal fluid, no intraretinal fluid, and no cystoid spaces at month 6
Time Frame: Month 0 to 6
Population: All participants with central subfield thickness recorded at Month 6
Measure: Number; unit: study eyes
Arm/Group | Aflibercept | Bevacizumab
Number analyzed (Participants) | 169 | 172
study eyes | 92 | 49

ADVERSE EVENTS:
Time Frame: Month 0 to 6
Arm/Group | Aflibercept | Bevacizumab
All-Cause Mortality (participants affected / at risk) | 1/180 | 1/182
Serious Adverse Events (participants affected / at risk) | 14/180 | 14/182
Other Adverse Events (participants affected / at risk) | 82/180 | 98/182
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Aflibercept (N=180) | Bevacizumab (N=182)
Acute kidney injury (Renal and urinary disorders) | 1 (1) | 0 (0)
Acute myocardial infarction (Cardiac disorders) | 0 (0) | 1 (1)
Acute respiratory failure (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Alcohol abuse (Psychiatric disorders) | 0 (0) | 1 (1)
Ankle fracture (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Arthritis (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Atrial fibrillation (Cardiac disorders) | 0 (0) | 1 (2)
Blood sodium decreased (Investigations) | 0 (0) | 1 (1)
Bronchitis (Infections and infestations) | 1 (1) | 0 (0)
Cardiac failure congestive (Cardiac disorders) | 1 (1) | 0 (0)
Cerebrovascular accident (Nervous system disorders) | 1 (1) | 0 (0)
Cerebrovascular stenosis (Nervous system disorders) | 0 (0) | 1 (1)
Chronic obstructive pulmonary disease (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Clostridium difficile colitis (Infections and infestations) | 0 (0) | 1 (1)
Dehydration (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
Diabetic foot infection (Infections and infestations) | 1 (1) | 0 (0)
Escherichia infection (Infections and infestations) | 1 (1) | 0 (0)
Gastrointestinal haemorrhage (Gastrointestinal disorders) | 0 (0) | 1 (1)
Hernia repair (Surgical and medical procedures) | 0 (0) | 1 (1)
Hypercoagulation (Blood and lymphatic system disorders) | 0 (0) | 1 (1)
Hypersensitivity (Immune system disorders) | 0 (0) | 1 (1)
Hypertension (Vascular disorders) | 1 (1) | 0 (0)
Hypertensive crisis (Vascular disorders) | 1 (1) | 0 (0)
Hypoglycaemia (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
Lymphoplasmacytoid lymphoma/immunocytoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Meningitis streptococcal (Infections and infestations) | 0 (0) | 1 (1)
Mental status changes (Psychiatric disorders) | 1 (1) | 0 (0)
Myocardial infarction (Cardiac disorders) | 1 (1) | 1 (1)
Neoplasm malignant (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Non-infectious endophthalmitis (Eye disorders) | 0 (0) | 1 (1)
Oesophageal adenocarcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Osteoarthritis (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Peripheral vascular disorder (Vascular disorders) | 1 (1) | 0 (0)
Pneumonia (Infections and infestations) | 0 (0) | 2 (2)
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Renal cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Sepsis (Infections and infestations) | 0 (0) | 1 (1)
Vertigo (Ear and labyrinth disorders) | 0 (0) | 1 (1)
Waldenstrom's macroglobulinaemia (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Aflibercept (N=180) | Bevacizumab (N=182)
Abdominal pain (Gastrointestinal disorders) | 0 (0) | 1 (1)
Acarodermatitis (Infections and infestations) | 0 (0) | 1 (1)
Acute kidney injury (Renal and urinary disorders) | 1 (1) | 2 (2)
Anaemia (Blood and lymphatic system disorders) | 1 (1) | 0 (0)
Aneurysm (Vascular disorders) | 0 (0) | 1 (1)
Angle closure glaucoma (Eye disorders) | 0 (0) | 2 (2)
Ankle fracture (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Anxiety (Psychiatric disorders) | 1 (1) | 1 (1)
Arteriovenous fistula aneurysm (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Arthralgia (Musculoskeletal and connective tissue disorders) | 3 (3) | 2 (2)
Asthenia (General disorders) | 0 (0) | 2 (2)
Atypical pneumonia (Infections and infestations) | 0 (0) | 1 (1)
Back pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 3 (3)
Bacterial infection (Infections and infestations) | 0 (0) | 1 (1)
Benign prostatic hyperplasia (Reproductive system and breast disorders) | 1 (1) | 0 (0)
Bladder cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Bladder neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Blepharitis (Eye disorders) | 0 (0) | 1 (1)
Blood cholesterol increased (Investigations) | 0 (0) | 1 (1)
Blood glucose increased (Investigations) | 0 (0) | 1 (1)
Blood pressure increased (Investigations) | 1 (1) | 3 (3)
Blood sodium decreased (Investigations) | 0 (0) | 1 (1)
Bradycardia (Cardiac disorders) | 0 (0) | 1 (1)
Bronchitis (Infections and infestations) | 4 (4) | 2 (2)
Bronchitis viral (Infections and infestations) | 1 (1) | 0 (0)
Cardiac failure congestive (Cardiac disorders) | 1 (1) | 0 (0)
Carpal tunnel syndrome (Nervous system disorders) | 0 (0) | 1 (1)
Cataract (Eye disorders) | 4 (4) | 2 (3)
Cataract nuclear (Eye disorders) | 0 (0) | 1 (1)
Cataract traumatic (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Catheter site haemorrhage (General disorders) | 0 (0) | 1 (1)
Cellulitis (Infections and infestations) | 1 (1) | 0 (0)
Cervical radiculopathy (Nervous system disorders) | 1 (1) | 0 (0)
Charles Bonnet syndrome (Eye disorders) | 1 (1) | 0 (0)
Chest pain (General disorders) | 3 (3) | 0 (0)
Chronic obstructive pulmonary disease (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Clostridium difficile colitis (Infections and infestations) | 1 (1) | 0 (0)
Clostridium difficile infection (Infections and infestations) | 0 (0) | 1 (1)
Conjunctival haemorrhage (Eye disorders) | 4 (4) | 14 (16)
Conjunctival hyperaemia (Eye disorders) | 1 (4) | 1 (1)
Conjunctival oedema (Eye disorders) | 0 (0) | 1 (1)
Constipation (Gastrointestinal disorders) | 1 (1) | 1 (1)
Contusion (Injury, poisoning and procedural complications) | 2 (2) | 0 (0)
Corneal abrasion (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Costochondritis (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Cough (Respiratory, thoracic and mediastinal disorders) | 3 (3) | 1 (1)
Cyst (General disorders) | 0 (0) | 1 (1)
Diabetes mellitus (Metabolism and nutrition disorders) | 1 (1) | 2 (2)
Diabetic retinopathy (Eye disorders) | 0 (0) | 1 (1)
Diverticulitis (Infections and infestations) | 1 (1) | 1 (1)
Dizziness (Nervous system disorders) | 2 (2) | 2 (3)
Drug hypersensitivity (Immune system disorders) | 0 (0) | 1 (1)
Dry eye (Eye disorders) | 1 (2) | 2 (3)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Endodontic procedure (Surgical and medical procedures) | 1 (1) | 0 (0)
Eye irritation (Eye disorders) | 3 (3) | 2 (3)
Eye pain (Eye disorders) | 6 (8) | 3 (3)
Eye pruritus (Eye disorders) | 1 (1) | 1 (1)
Eye swelling (Eye disorders) | 0 (0) | 2 (2)
Eyelid disorder (Eye disorders) | 0 (0) | 1 (1)
Eyelid pain (Eye disorders) | 1 (1) | 0 (0)
Facial pain (General disorders) | 1 (1) | 0 (0)
Fall (Injury, poisoning and procedural complications) | 2 (2) | 5 (5)
Foreign body sensation in eyes (Eye disorders) | 1 (3) | 1 (1)
Gastroenteritis viral (Infections and infestations) | 2 (2) | 0 (0)
Gingivitis (Infections and infestations) | 1 (1) | 0 (0)
Glaucoma (Eye disorders) | 0 (0) | 1 (1)
Gout (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
Haematochezia (Gastrointestinal disorders) | 1 (1) | 0 (0)
Haematoma (Vascular disorders) | 1 (1) | 0 (0)
Haematoma infection (Infections and infestations) | 1 (1) | 0 (0)
Haematuria (Renal and urinary disorders) | 0 (0) | 1 (1)
Headache (Nervous system disorders) | 2 (2) | 6 (6)
Herpes zoster (Infections and infestations) | 1 (1) | 0 (0)
Hypersensitivity (Immune system disorders) | 0 (0) | 1 (1)
Hypertension (Vascular disorders) | 3 (3) | 5 (5)
Hypertriglyceridaemia (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
Hypoglycaemia (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
Hypothyroidism (Endocrine disorders) | 1 (1) | 0 (0)
Influenza (Infections and infestations) | 1 (1) | 1 (1)
Intraocular pressure increased (Investigations) | 1 (2) | 5 (5)
Joint injury (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Joint swelling (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Keratopathy (Eye disorders) | 1 (1) | 0 (0)
Lacrimation increased (Eye disorders) | 1 (1) | 1 (2)
Large intestine polyp (Gastrointestinal disorders) | 1 (1) | 0 (0)
Ligament sprain (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Localised infection (Infections and infestations) | 1 (1) | 0 (0)
Macular hole (Eye disorders) | 1 (1) | 0 (0)
Macular ischaemia (Eye disorders) | 0 (0) | 1 (1)
Macular oedema (Eye disorders) | 0 (0) | 1 (1)
Maculopathy (Eye disorders) | 1 (1) | 0 (0)
Metabolic encephalopathy (Nervous system disorders) | 0 (0) | 1 (1)
Metamorphopsia (Eye disorders) | 0 (0) | 1 (1)
Migraine (Nervous system disorders) | 0 (0) | 1 (1)
Muscle spasms (Musculoskeletal and connective tissue disorders) | 0 (0) | 2 (2)
Muscular weakness (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Musculoskeletal stiffness (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Myalgia (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Myocardial infarction (Cardiac disorders) | 1 (1) | 0 (0)
Nasopharyngitis (Infections and infestations) | 3 (3) | 6 (6)
Nausea (Gastrointestinal disorders) | 2 (2) | 1 (1)
Neuralgia (Nervous system disorders) | 0 (0) | 1 (1)
Ocular discomfort (Eye disorders) | 0 (0) | 1 (1)
Ocular hyperaemia (Eye disorders) | 0 (0) | 1 (1)
Ocular hypertension (Eye disorders) | 1 (2) | 1 (1)
Ophthalmoplegia (Eye disorders) | 0 (0) | 1 (1)
Optic disc hyperaemia (Eye disorders) | 0 (0) | 1 (1)
Optic neuritis (Nervous system disorders) | 0 (0) | 1 (1)
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 1 (1)
Osteoarthritis (Musculoskeletal and connective tissue disorders) | 0 (0) | 2 (2)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 0 (0) | 2 (2)
Papilloedema (Eye disorders) | 0 (0) | 1 (1)
Paranasal sinus discomfort (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Parkinson's disease (Nervous system disorders) | 1 (1) | 0 (0)
Periorbital haemorrhage (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Peripheral nerve decompression (Surgical and medical procedures) | 0 (0) | 1 (1)
Pharyngitis streptococcal (Infections and infestations) | 0 (0) | 1 (1)
Photophobia (Eye disorders) | 1 (1) | 1 (2)
Photopsia (Eye disorders) | 0 (0) | 1 (1)
Plantar fasciitis (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Pneumonia (Infections and infestations) | 1 (1) | 0 (0)
Polyneuropathy (Nervous system disorders) | 0 (0) | 1 (1)
Posterior capsule opacification (Eye disorders) | 0 (0) | 1 (1)
Procedural pain (Injury, poisoning and procedural complications) | 1 (1) | 1 (1)
Prostatomegaly (Reproductive system and breast disorders) | 0 (0) | 2 (2)
Pruritus (Skin and subcutaneous tissue disorders) | 0 (0) | 2 (2)
Pulmonary hypertension (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Pyrexia (General disorders) | 0 (0) | 2 (2)
Rash pruritic (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
Respiratory tract congestion (Infections and infestations) | 1 (1) | 0 (0)
Respiratory tract infection (Infections and infestations) | 0 (0) | 2 (2)
Retinal collateral vessels (Eye disorders) | 0 (0) | 1 (1)
Retinal exudates (Eye disorders) | 2 (2) | 3 (3)
Retinal haemorrhage (Eye disorders) | 0 (0) | 3 (3)
Retinal vascular disorder (Eye disorders) | 0 (0) | 1 (1)
Retinal vein occlusion (Eye disorders) | 2 (2) | 2 (2)
Rotator cuff syndrome (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Sarcoidosis (Immune system disorders) | 0 (0) | 1 (1)
Sciatica (Nervous system disorders) | 1 (1) | 1 (1)
Seasonal allergy (Immune system disorders) | 3 (3) | 0 (0)
Sinusitis (Infections and infestations) | 2 (2) | 5 (5)
Sleep apnoea syndrome (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Squamous cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Stomatitis (Gastrointestinal disorders) | 1 (1) | 0 (0)
Subretinal fluid (Eye disorders) | 1 (1) | 0 (0)
Syncope (Nervous system disorders) | 0 (0) | 2 (2)
Temporomandibular joint syndrome (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Tendon injury (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Tinea pedis (Infections and infestations) | 0 (0) | 1 (1)
Tooth extraction (Surgical and medical procedures) | 0 (0) | 1 (1)
Tooth fracture (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Tooth infection (Infections and infestations) | 1 (1) | 0 (0)
Tremor (Nervous system disorders) | 0 (0) | 1 (1)
Upper respiratory tract infection (Infections and infestations) | 2 (2) | 2 (2)
Urinary retention (Renal and urinary disorders) | 0 (0) | 1 (1)
Urinary tract infection (Infections and infestations) | 3 (3) | 6 (6)
Urticaria (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
Vertigo (Ear and labyrinth disorders) | 1 (1) | 0 (0)
Vertigo positional (Ear and labyrinth disorders) | 1 (1) | 0 (0)
Vision blurred (Eye disorders) | 1 (1) | 5 (8)
Visual acuity reduced (Eye disorders) | 3 (4) | 7 (7)
Visual impairment (Eye disorders) | 1 (1) | 0 (0)
Vitreous adhesions (Eye disorders) | 1 (1) | 0 (0)
Vitreous detachment (Eye disorders) | 6 (6) | 3 (3)
Vitreous floaters (Eye disorders) | 6 (6) | 8 (8)
Vitreous opacities (Eye disorders) | 0 (0) | 1 (1)
Vomiting (Gastrointestinal disorders) | 0 (0) | 1 (1)
Vulva cyst (Reproductive system and breast disorders) | 0 (0) | 1 (1)
Wound (Injury, poisoning and procedural complications) | 1 (1) | 1 (1)
Wrist fracture (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Trial results can not be discussed until they have been made available to the public.